CLINICAL TRIAL: NCT00005989
Title: A Phase II Study of Farnesyl Transferase Inhibitor R115777 in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: R115777 in Treating Patients With Recurrent or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Julian R. Molina, M.D., Ph.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000067978; U01CA069912 (NIH); P30CA015083 (NIH); 982401 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2000-07-05; First posted 2004-04-20 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tipifarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of R115777 in treating patients who have recurrent or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the response rate of patients with recurrent or metastatic non-small cell lung cancer when treated with tipifarnib.
* Determine the clinical toxicities of this treatment in these patients.
* Assess the overall survival and time to progression of this patient population when treated with this regimen.
* Evaluate the inhibition of protein farnesylation in vivo and correlate such inhibition to plasma levels of tipifarnib.
* Evaluate the occurrence of CYP450 polymorphisms and relate these to drug toxicity, pharmacokinetics, and response to this treatment in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed recurrent or metastatic non-small cell lung cancer (NSCLC)
* Measurable disease

  * At least 20 mm in at least one dimension
  * Nonmeasurable is defined as any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN (no greater than 5 times ULN in case of hepatic metastases)

Renal

* Creatinine no greater than 2 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other prior malignancy in past 5 years except adequately treated basal cell or squamous cell skin cancer or other adequately treated noninvasive carcinomas
* No other concurrent severe underlying disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic, gene, or immunotherapy

Chemotherapy

* No prior chemotherapy for NSCLC except low dose cisplatin as radiosensitizer

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy to less than 25% of bone marrow allowed

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, MD, Study Chair — Mayo Clinic; Elizabeth Johnson, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota